CLINICAL TRIAL: NCT05890274
Title: Improving Outpatient Comprehensive Atrial Fibrillation Care Across Central North Carolina Through Direct Primary Care and Patient Engagement
Brief Title: Atrial Fibrillation (AF) and Electrocardiogram (EKG) Interpretation Project ECHO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); Wake Forest University (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-1350a
Record Dates: First submitted 2023-05-17; First posted 2023-06-06 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AF and EKG Interpretation Project ECHO (Experimental): All recruited participants participate in the AF and EKG Interpretation Project ECHO educational intervention.
  Interventions: Other: AF and EKG Interpretation Project ECHO

INTERVENTIONS:
Other: AF and EKG Interpretation Project ECHO — The AF and EKG Interpretation Project ECHO program is delivered via Zoom videoconferencing technology and includes 12, 1-hour long sessions that involve education on best practice management of AF for primary care providers. Each session includes an EKG challenge, case presentation by a participant, didactic presentation, and time for open Q&A. Supplementary materials are made available to all participants.

SUMMARY:
The goal of this study is to determine the effectiveness of a direct-to-provider virtual education program ("AF and EKG Interpretation Project ECHO") for primary care providers who manage patients with atrial fibrillation (AF). The main questions this study aims to answer are:

1. Will participants have improvement in knowledge and confidence in managing patients with atrial fibrillation after program completion?
2. Will quality and performance metrics improve at the patient level for program participants?

Participants will be asked to:

* Participate in 12 hours of virtual education sessions over twelve weeks via Zoom.
* Complete a knowledge and confidence assessment online before the program starts and after its completion.

ELIGIBILITY:
Inclusion Criteria:

* Primary care provider (Physician, Nurse Practitioner, Physician Assistant) with primary practice in the state of North Carolina
* Care for adult population

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in Number of Patients Prescribed Appropriate Anticoagulation | 1-year prior to intervention session 1 and 1-year post intervention session 12
  This outcome measures the number of patients prescribed appropriate anticoagulation medication based on risk factors for stroke including congestive heart failure (C), hypertension (H), Age >74 (A2), Diabetes (D), prior stroke or transient ischemic attack (TIA) (S2), vascular disease (V), age 65-74 (A), female sex (Sc), commonly referred to as CHA2DS2-VASc stroke risk score for patients with atrial fibrillation. CHA2DS2-VASc score includes 7 indicators of stroke risk (age (<65=0, 65-74=1, 75+= 2), sex (male=0, female=1), heart failure (no=0, yes=1), hypertension (no=0, yes=1), prior stroke/TIA (no=0, yes=2), history of vascular disease (no=0, yes=1), and diabetes (no=0, yes=1). Anticoagulation is indicated for a female with a score 3 or higher and males with a score of 2 or higher. This information will be collected from electronic health records of patients cared for by providers who participated in the program.

SECONDARY OUTCOMES:
Change Score on Provider Knowledge Assessment | Baseline and 12 weeks post intervention session 12
  This outcome measures the change in provider knowledge in Afib management using an internally developed knowledge test. The test includes 25 multiple choice questions based on clinical case scenarios. The number of questions answered correctly prior to the start of the program will be compared with the number of questions answered correctly after program completion.
Change in Provider Confidence Level | Baseline and 12 weeks post intervention session 12
  This outcome measures the change in provider confidence in managing patients with Afib. Confidence is measured using an internally developed confidence scale on 9 key areas of management related to Afib. Each of the 9 questions is measured on a 5 point likert scale from 1 (not at all confident) to 5 (extremely confident) for a total score ranging from 9 to 45 with the higher the score related to higher confidence in managing patients with Afib.
Change in Number of Patients Prescribed Appropriate Antiplatelet Therapy | 1-year prior to intervention session 1 and 1-year post intervention session 12
  This outcome measures the number of Afib patients prescribed appropriate antiplatelet therapy. Antiplatelet therapy is considered appropriate if the patient has a history of vascular disease. Antiplatelet therapy will be considered not appropriate if the patient has a history of Afib and no history of vascular disease. This information will be collected from electronic health records of patients cared for by providers who participated in the program.
Change in Number of Patients with Blood Pressure at Goal | 1-year prior to intervention session 1 and 1-year post intervention session 12
  This outcome measures the number of patients who achieve blood pressure at goal at outpatient primary care visits. Blood pressure at goal is determined by guidelines set forth by the American College of Cardiology (ACC) and American Heart Association (AHA) which is less than 130 mmHg systolic and less than 80 mmHg diastolic. This information will be collected from electronic health records of patients cared for by providers who participated in the program.
Change in Number of Patients with Heart Rate at Target | 1-year prior to intervention session 1 and 1-year post intervention session 12
  This outcome measures the number of patients who achieve heart rate at goal at outpatient primary care visits. Heart rate at goal is determined by guidelines set forth by the American Heart Association (AHA) and American College of Cardiology (ACC) which recommends a heart rate of less than 110 beats per minute. This information will be collected from electronic health records of patients cared for by providers who participated in the program.
Change in Number of Emergency Department Visits or Hospitalizations for AF or Stroke | 1-year prior to intervention session 1 and 1-year post intervention session 12
  This outcome measures the number of patient visits to the emergency department and number of hospitalizations for a primary diagnosis of Afib or stroke. The number of visits 1 year prior to the intervention will be compared to the number of visits during the 1 year following intervention session 12. This information will be collected from electronic health records of patients cared for by providers who participated in the program.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gehi, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society in Collaboration With the Society of Thoracic Surgeons. Circulation. 2019 Jul 9;140(2):e125-e151. doi: 10.1161/CIR.0000000000000665. Epub 2019 Jan 28. No abstract available. PMID 30686041
- [Background] Carey RM, Wright JT Jr, Taler SJ, Whelton PK. Guideline-Driven Management of Hypertension: An Evidence-Based Update. Circ Res. 2021 Apr 2;128(7):827-846. doi: 10.1161/CIRCRESAHA.121.318083. Epub 2021 Apr 1. PMID 33793326
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- See also: University of New Mexico Project ECHO Website — https://hsc.unm.edu/echo/